CLINICAL TRIAL: NCT06697535
Title: Efficacy and Safety of JYP0061 in Patients With Acute Neuromyelitis Spectrum Disease (NMOSD): a Multicenter, Randomized, Open-label, Positive-controlled, Two-stage Exploratory Phase 2 Trial
Brief Title: A Study to Evaluate the Efficacy and Safety of JYP0061 in Patients With Acute Neuromyelitis Spectrum Disease (NMOSD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYP0061M202
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Methylprednisolone; Glucocorticoids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose JYP0061 + Reduced Dose Glucocorticoids (Group A) (Experimental): Participants in this group will receive JYP0061, starting with a higher dose for the initial weeks, followed by a reduced maintenance dose. In addition, participants will receive a regimen of glucocorticoids, starting with intravenous administration and transitioning to oral dosing with a gradually tapering dose over time.
  Interventions: Drug: JYP0061; Drug: Intravenous Glucocorticoids; Drug: Oral Glucocorticoids
- Standard Dose Glucocorticoids (Groups B1 and B2) (Active Comparator): Participants in this group will receive a standard glucocorticoid regimen, starting with intravenous glucocorticoids at higher doses, with doses tapering over time, and then transitioning to an oral glucocorticoid regimen that also tapers gradually. During the second phase, adjustments may be made based on the participant's clinical response.
  Interventions: Drug: Intravenous Glucocorticoids; Drug: Oral Glucocorticoids
- High-dose JYP0061 (Group C) (Experimental): Participants in this group will receive a higher dose of JYP0061 for the initial weeks, followed by a lower maintenance dose for the remainder of the study period.
  Interventions: Drug: JYP0061

INTERVENTIONS:
Drug: JYP0061 — Administered orally with a dose reduction over time as specified in Arm descriptions. Tablets are taken within a specific time frame after meals.
  Other Names: Experimental Drug Group
  Arms: High-dose JYP0061 (Group C); Low-dose JYP0061 + Reduced Dose Glucocorticoids (Group A)
Drug: Intravenous Glucocorticoids — Administered intravenously with a gradually decreasing dose over time, as specified in the Standard Dose Glucocorticoids arm.
  Other Names: Methylprednisolone
  Arms: Low-dose JYP0061 + Reduced Dose Glucocorticoids (Group A); Standard Dose Glucocorticoids (Groups B1 and B2)
Drug: Oral Glucocorticoids — Administered orally with a tapered dosing schedule, as specified in the Standard Dose Glucocorticoids arm, with adjustments based on participant response.
  Other Names: Prednisone
  Arms: Low-dose JYP0061 + Reduced Dose Glucocorticoids (Group A); Standard Dose Glucocorticoids (Groups B1 and B2)

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety, of JYP0061 in acute NMOSD patients. The main questions it aims to answer are: efficacy and safety of JYP0061 in acute NMOSD patients. Participants will be treated with low-dose JYP0061 in combination with reduced dose glucocorticoids or standard dose glucocorticoids or high-dose JYP0061. Efficacy and safety evaluations will be conducted according to the protocol.

DETAILED DESCRIPTION:
This study will be an open-label, multicenter phase 2 clinical trial. After being informed about the study and potential risks, all subjects giving written informed consent will undergo a 2-week screening period to determine eligibility for study entry. And then subjects will be treated with low-dose JYP0061 in combination with reduced dose glucocorticoids or standard dose glucocorticoids. The efficacy and safety measures will be conducted according to the protocol. If JYP0061 is effective and safe for acute NMOSD patients, then subjects will be treated with high-dose JYP0061 or standard dose glucocorticoid. The efficacy and safety measures will be conducted according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Neuromyelitis spectrum disease (NMOSD) patients according to 2015 International consensus diagnostic criteria.
* Positive Aquaporin 4 immunoglobulin G (AQP4-IgG)
* Patients with acute NMOSD
* Female serum pregnancy test results were negative at the time of screening, subject (including partner) had no child-rearing plan and voluntarily adopted double contraceptive (non-oral contraceptives) within 6 months from screening to the last study drug administration, and had no sperm/egg donation plan;
* Have fully understood this study, voluntarily participate in the experiment, and voluntarily sign the written informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* Suspected or clear allergy to similar ingredients or any ingredient in the study drug, or allergic constitution;
* Symptoms improved in the acute phase before the study drug was used;
* Unable to complete MRI or gadolinium enhanced examination;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving clinical recovery based on EDSS after 6 weeks of treatment | 6 weeks after the first administration of the medication.
  This outcome assesses the clinical efficacy of JYP0061 in acute-phase NMOSD patients. The proportion of participants achieving various levels of recovery-Complete Recovery (CR), Good Recovery (GR), Moderate Recovery (MR), and Poor Recovery (PR)-will be evaluated based on the Expanded Disability Status Scale (EDSS) after 6 weeks of treatment.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JYP0061 in NMOSD Participants | Weeks 2, 4, 6, 14, and 26.
  This outcome measures the maximum plasma concentration (Cmax) of JYP0061 in participants with NMOSD, assessed at Weeks 2, 4, 6, 14, and 26 following administration.
Apparent Clearance (CL/F) of JYP0061 in NMOSD Participants | Weeks 2, 4, 6, 14, and 26.
  This outcome measures the apparent clearance (CL/F) of JYP0061 in participants with NMOSD, assessed at Weeks 2, 4, 6, 14, and 26 following administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital，Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No